CLINICAL TRIAL: NCT01156831
Title: Consequences of Positron-Emission-Tomography/Computed Tomography (PET/CT) Based Radiotherapy Treatment Planning for Clinical Outcome in Esophageal Cancer Patients
Brief Title: PET-CT Based Radiotherapy in Esophageal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 09-18-12/08
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal cancer; PET-CT planning
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the locoregional control in PET/CT based radiotherapy treatment planning in the treatment of esophageal cancer patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine the locoregional control in PET/CT based radiotherapy treatment planning in the treatment of esophageal cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma or squamous cell carcinoma of the esophagus
* Local curable disease able to undergo Chemoradiotherapy.

Exclusion Criteria:

* Metastasized disease.
* Previous or concurrent malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Locoregional control | 2 years and 5 years

SECONDARY OUTCOMES:
Overall Survival | 2 years and 5 years
Disease Free survival | 2 years and 5 years
Tumor regression grade | At the time of surgery
  Tumor regression grade at time of surgery evaluated by pathologist.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Lammering, MD PhD, Principal Investigator — Radiation Oncology, Maastro Clinic; Meindert Sosef, MD PhD, Principal Investigator — Atrium Hospital Heerlen
Locations (5):
- Netherlands (5):
  - Atrium Hospital, Heerlen
  - University Medical Center, Maastricht
  - St. Laurentius Hospital, Roermond
  - Maasland Hospital, Sittard
  - St. Jansgasthuis, Weert